CLINICAL TRIAL: NCT00904800
Title: A Single-blind, Randomised, Placebo-controlled, Parallel-group, Single Centre Phase I Study to Assess the Safety, Tolerability and Pharmacokinetics of Extended-release Tablets AZD0837 After Single and Repeated Oral Administration to Young Healthy Male Japanese Subjects
Brief Title: AZD0837 Extended Release (ER) Japan Study
Acronym: ER J ph I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Wahlander Karin, MD, PhDMedical Science Director, AstraZeneca R&D Molndal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D1250C00055
Record Dates: First submitted 2009-05-13; First posted 2009-05-20 (Estimated); Last update posted 2009-07-13 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
Keywords: Phase I; Healthy volunteers
MeSH Terms: interventions — AZD 0837

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Low dose
  Interventions: Drug: AZD0837
- 2 (Experimental): Middle dose
  Interventions: Drug: AZD0837
- 3 (Experimental): High dose
  Interventions: Drug: AZD0837
- 4 (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD0837 — tablet, oral, once daily, 1+5 days
  Arms: 1; 2; 3
Drug: Placebo — Placebo
  Arms: 4

SUMMARY:
This phase I study will evaluate safety and tolerability after repeated doses of AZD0837.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male Japanese subject aged between 20 to 45 years inclusive

Exclusion Criteria:

* Acute illness (including ongoing or history of liver disease), trauma or surgical procedures within two weeks before Visit 1 or pre first dose in Visit 2
* Intake of another investigational drug within 4 months before Visit 1 or pre first dose in Visit 2
* Blood donation and/or sampling in excess of 200 mL of whole blood within the preceding 4 weeks, 400 mL of whole blood within the preceding 12 weeks and/or 1200 mL of whole blood within the preceding 12 months, before Visit 1 or pre first dose in Visit 2

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2009-05; Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of AZD0837 after single and repeated oral dosing of AZD0837 extended release (ER) tablet, in Japanese healthy subjects. | All assessments are made at each visit, at least daily, during the study.

SECONDARY OUTCOMES:
To investigate the pharmacokinetics (PK) of AZD0837, AR H069927XX and AR-H067637XX after single and repeated oral dosing of AZD0837 ER tablet, in Japanese healthy subjects. | Blood samples will be taken before and after study drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroyuki Fukase, MD, PhD, Principal Investigator — CPC Clinic, Medipolis Medical Research Institute, Kagoshima, Japan
Locations (1):
- Research Site, Kagoshima, Japan